CLINICAL TRIAL: NCT03322319
Title: acTive scrEening of cArdiac aMyloidosis in the Caribbean's
Brief Title: Frequency of Cardiac Amyloidosis in the Caribbean's. (TEAM Amylose)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12/B/17
Record Dates: First submitted 2017-10-23; First posted 2017-10-26 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Left Ventricular Hypertrophy
Keywords: Cardiac amyloidosis; Caribbean; Diagnosis; Transthyretin
MeSH Terms: conditions — Hypertrophy, Left Ventricular; Amyloid Neuropathies, Familial; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- left Ventricular Hypertrophy (Experimental): Patients with left ventricular wall thickness measuring 15mm or more, or patients with a suggestive left ventricular echogenicity. Procedure/surgery will be performed following a diagnostic tree.
  Interventions: Procedure: Tissue biopsies

INTERVENTIONS:
Procedure: Tissue biopsies — It is commonly accepted that the diagnosis of cardiac amyloidosis may be based on presence of characteristic cardiac abnormalities in echography, associated with the detection of bi-refractive appearance deposits in polarized light after congo red staining of a biopsy fragment.
  Usually a biopsy of the abdominal fat or salivary glands can suffice. More rarely, in case of persistent doubt (eg negativity of congo red despite a characteristic appearance, which may occur in 20 to 30% of cases), it will be necessary to perform an endomyocardial biopsy (EMB).

SUMMARY:
The frequency of cardiac amyloidosis among patients presenting with a so-called left ventricular hypertrophy remains unknown. This problem is especially relevant in the Caribbean's, where an amyloidosis-prone mutation of transthyretin gene might be frequent.

DETAILED DESCRIPTION:
Cardiac amyloidosis is a very poorly known disease, in its frequency, its mechanisms, its treatment. This lack of knowledge is a major limitation to the improvement, indispensable, of the care of the patients. In clinical routine, particularly in West Indies-Guyana, cardiac amyloidosis is a disease poorly identified, whose management remains to be optimized. Concordant observations suggest that the frequency of the disease could be significant in the Antilles-Guyana: aging of the population, high frequency of an amyloidogenic mutation (Val122Il mutation of the transthyretin gene) found in 4% of the Afro-American population, recent identification in Martinique by a neurology team of a new founding mutation of the transthyretin gene that may cause the disease.

These elements justified the setting up of a multidisciplinary group whose objective is to contribute to the improvement of screening, treatment, and follow-up of patients with cardiac amyloidosis.

An identical diagnostic algorithm will be followed in all centers. Therapeutic management will be left to the discretion of the health care teams, who will be communicated regularly, the latest management recommendations.

A frequency of 30% is expected and will be assessed with a power of 80% and an alpha risk of 0.05. Quantitative and qualitative data will be described as usual. Differences between groups will be assessed with parametric or non-parametric tests.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years,
* Residency in French Caribbean Regions
* Access to healthcare coverage,
* Written informed consent obtained

Exclusion Criteria:

* Evidence of another cause for left ventricular hypertrophy (uncontrolled severe high blood pressure, untreated severe aortic stenosis, family history of hypertrophic cardiomyopathy)
* Inability to deliver informed consent,
* Presence of a known severe disease impending participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2013-09-23 (Actual); Primary Completion 2015-12-02 (Actual); Study Completion 2016-01-18 (Actual)

PRIMARY OUTCOMES:
Diagnosis of cardiac amyloidosis. | 3 months
  Diagnosis procedures involve clinical exam, echocardiography, MRI, SPECT, tissue biopsies, and will be realized following a diagnostic tree.

SECONDARY OUTCOMES:
Subtyping of cardiac amyloidosis | 2 years
  To refine the genetic epidemiology of cardiac amyloidosis in the Caribbean's

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyn INAMO, MD-PhD, Principal Investigator — Centre Hospitalier Universitaire de Martinique, France
Locations (2):
- Centre Hospitalier de Basse-Terre, Basse-Terre, Guadeloupe
- CHU de Martinique, La Trinité, Martinique

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After the main publication of the results, for not limited time.
Access Criteria: The conditions for the transfer of all or part of the database of the research are decided by the investigator coordinator / sponsor of the research and are the subject of a written contract.

REFERENCES:
- [Result] Oliveira Da Silva L, Fabre J, Monfort A, Villeret J, Citony I, Cohen-Tenoudji P, Lebbadi M, Martin D, Molinie V, Inamo J. 'Green Apple' Heart Failure. West Indian Med J. 2014 Jul 3;63(6):673-5. doi: 10.7727/wimj.2013.255. Epub 2014 Jun 25. PMID 25803389